CLINICAL TRIAL: NCT05051891
Title: A Randomized, Open-label, Multi-center, Phase III Study of Orelabrutinib in Combination With Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) vs. R-CHOP Alone in Patients With Treatment-naїve Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00113
Record Dates: First submitted 2021-09-15; First posted 2021-09-21 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-08

CONDITIONS: Treatment-naїve Mantle Cell Lymphoma
MeSH Terms: interventions — orelabrutinib; R-CHOP protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental): Orelabrutinib in Combinaion with Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP)
  Interventions: Drug: Orelabrutinib and R-CHOP
- The control group (Experimental): R-CHOP
  Interventions: Drug: R-CHOP

INTERVENTIONS:
Drug: Orelabrutinib and R-CHOP — Orelabrutinib in Combinaion with Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP)
  Arms: the experimental group
Drug: R-CHOP — Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP)
  Arms: The control group

SUMMARY:
To evaluate the efficacy of orelabrutinib combined with R-CHOP vs. R-CHOP alone in the treatment of treatment-naїve mantle cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. 65 < age <80, or 60 ≤ age ≤65 and is ineligible for autologous stem cell transplantation as assessed by the investigator
2. Histopathological confirmed MCL and either expression of cyclin D1 or t (11;14) chromosomal translocation (in association with CD20). The verification will be based on central review of the local pathology report.
3. No previous systemic treatment for MCL.
4. ECOG physical strength score is 0-2.
5. Expected survival time >6 months.
6. Voluntary written informed consent prior to screening.

Exclusion Criteria:

1. Uncontrolled or significant cardiovascular diseases
2. History of stroke or intracranial hemorrhage within 6 months before first administration of study treatment.
3. Any mental or cognitive impairments which may limit the subject 's understanding and execution of informed consent as well as study compliance;
4. Pregnant or breastfeeding women and those who do not agree to take contraceptive measures.
5. Conditions in which a potentially life-threatening illness or severe organ dysfunction is not considered appropriate by the investigator.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 6 years
  To evaluate the Progression-free Survival (PFS) by the Independent Review Committee (IRC) according to the 2014 International Working Group Criteria for Non-Hodgkin Lymphoma (iwNHL).

SECONDARY OUTCOMES:
ORR | Up to 6 years
  Objective Response Rate
CRR | Up to 6 years
  Complete Response Rate
OS | Up to 6 years
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Anhui Province Cancer Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Tumor in Hunan Province, Hunan, Changsha
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Tumor Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaojing
  - The First Affiliated Hospital of Guangxi Medical University, Guangxi, Nanning
  - Shandong Provincial Hospital, Jinan, Shandong
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - he First Affiliated Hospital of Zhengjiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang